CLINICAL TRIAL: NCT03151525
Title: Comparison Between Two Therapeutic Strategies for the Maintenance of Clinical and Endoscopic Remission in Patients With Ulcerative Colitis Treated by Infliximab
Brief Title: Two Therapeutic Strategies for the Maintenance of Remission in Patients With Ulcerative Colitis
Acronym: SCILLA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1685
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Azathioprine; Infliximab

STUDY DESIGN:
Intervention Model Description: Randomized parallel two-arm prospective open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azathioprine (Experimental): Azathioprine 2-2.5 mg/kg/day, according to approved indication
  Interventions: Drug: Azathioprine
- Infliximab (Active Comparator): Infliximab 5 mg/kg every 8 weeks
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Azathioprine — AZA treatment after IFX withdrawal for maintenance of remission
  Arms: Azathioprine
Drug: Infliximab — IFX treatment for maintenance of remission
  Arms: Infliximab

SUMMARY:
Ulcerative colitis patients treated with Infliximab (IFX) in deep remission after at least 12 months of treatment will be randomized to continue IFX or to stop IFX and start Azathioprine (AZA).

Each patient will be followed for 12 months.

DETAILED DESCRIPTION:
All eligible subjects will be able to participate in the study at any infusion occurred after 12 months since the beginning. They will be screened by medical history, physical examination, blood and faecal tests (included C-reactive protein and faecal calprotectin), as required by clinical practice. No children, pregnant or breastfeeding women, or elder subjects will be included. A colonoscopy + biopsies in the area of greater inflammation will be performed within ± 3 weeks since the baseline visit. The subjects can then be randomized and receive their first dose of study medication.

Subjects will be then evaluated every 8 weeks for the following 12 months from the randomization. Clinical and blood tests will be performed, and the partial Mayo Score will be calculated at each visit, until the final visit, when a new colonoscopy with biopsies will be repeated and the global Mayo Score will be evaluated. At final visit a new faecal sample for calprotectin will be collected.

Safety of the study treatments will be evaluated at each study visit. In case of study agent discontinuation, the patient will be managed according to usual practice and followed for the entire study period. Patients randomized in AZA arm, could restart IFX.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -65 years
* Written informed consent and willing to adhere to study procedures.
* Therapy with infliximab since at least 12 months, with one infusion every 8 weeks (a maximum interval between two infusions of ± 3 weeks is allowed)
* Sustained steroid-free remission in the last 6 months prior to inclusion, except for use of steroids as a preventive measure for infliximab infusion reaction, if required by local guidelines.
* Global Mayo score at baseline ≤ 2
* All Mayo subscores ≤ 1
* Absence of rectal bleeding
* Effective methods to avoid pregnancy during the study period

Exclusion Criteria:

* Disabling and persisting extraintestinal manifestation at baseline
* Patients unable to comply with study procedures
* Known intolerance or previous allergic reaction to thiopurines
* Concomitant therapy with allopurinol
* Any disease not compatible with the use of infliximab or azathioprine, as per clinician's judgement.
* Need for dose escalation of infliximab in the last 12 months prior to baseline.
* White blood cell count < 3000/mmc or absolute clinically relevant lymphopenia at baseline
* Active pregnancy or breastfeeding; willing for pregnancy during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-10-03 (Estimated); Study Completion 2020-04-03 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 12 months
  relapse rate in the two study groups.

SECONDARY OUTCOMES:
Relapse time | 12 months
  Mean time to relapse in the two groups
Number of adverse events [Safety and Tolerability] | 12 months
  Number of adverse events of the two study strategies
Number of serious adverse events [Safety and Tolerability] | 12 months
  Number of serious adverse events of the two study strategies
Identification of potential risk factors for relapse. Age, sex, smoking habits, histological healing of mucosa and each Mayo subscore at baseline will be examined | 12 months
  Potential risk factor for relapse will be evaluated by univariable analysis, and a multivariable analysis will be performed for all factors with p<0.30. Risk factors will be also analysed by logistic regression. Analysis of predetermined baseline characteristics (age, sex, smoking habits, histological healing of mucosa at baseline, and each Mayo subscore (stool number, presence of blood, colonic ulcerations) excluding the physician global assessment) to identify predictive factors for relapse.

OTHER OUTCOMES:
Direct costs [Pharmacokinetics] | 12 months
  Direct costs of the two treatment strategies

CONTACTS AND LOCATIONS:
Locations (1):
- IBD Center, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523